CLINICAL TRIAL: NCT03653481
Title: Safety and Feasibility of Oligofructose-Enriched Inulin in Pediatric Inflammatory Bowel Disease
Brief Title: Treating IBD With Inulin
Acronym: TII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Beneo GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18-015331
Record Dates: First submitted 2018-08-28; First posted 2018-08-31 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Inflammatory Bowel Diseases
Keywords: diet; inulin; prebiotic; IBD; Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inulin (Experimental): Oligofructose-enriched Inulin (OI) administered for 8 weeks
  Interventions: Dietary Supplement: Oligofructose-enriched Inulin OI
- Placebo (Placebo Comparator): Maltodextrin placebo administered for 8 weeks
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Oligofructose-enriched Inulin OI — Consumed as a powder, 8g/d for children <50kg and 16g/d for children ≥50kg, divided in 2 daily doses.
  Other Names: Orafti®Synergy1
  Arms: Inulin
Dietary Supplement: Maltodextrin — Consumed as a powder, 8g/d for children <50kg and 16g/d for children ≥50kg, divided in 2 daily doses.
  Arms: Placebo

SUMMARY:
The purpose of this study is to see how the prebiotic inulin changes the gut bacteria (microbiome) of children and young adults with IBD and determine if this dietary intervention can help reduce disease activity.

DETAILED DESCRIPTION:
The pathogenesis of inflammatory bowel disease (IBD) is thought to be due to a combination of genetic, environmental and immunological factors. From a clinical stand point, there is great interest in determining if manipulation of the gut microbiota may be a viable therapeutic strategy in IBD patients. One such strategy involves the use of prebiotic. Prebiotics are oligosaccharides that cannot be enzymatically hydrolyzed in the small intestine, however serve as substrates for fermentation by commensal bacteria in the colon.

Investigators propose to evaluate the modulatory effects of the prebiotic inulin on the composition and function of the microbiota of children with IBD and determine the efficacy of this dietary intervention in reducing disease activity.

ELIGIBILITY:
Inclusion Criteria

* Males or females age 8-21 years.
* Parental/guardian permission (informed consent) and child assent.
* Pediatric diagnosis of inflammatory colonic or ileocolonic Crohn's disease (CD), ulcerative colitis (UC) or inflammatory bowel disease-unclassified (IBDU), as defined by endoscopy, radiology, and clinical findings.
* Clinical disease activity index compatible with:

  * For patients with CD:

    * Pediatric Crohn's Disease Activity Index (PCDAI) ≤15 or short PCDAI (sPCDAI) ≤17.5 (if unable to complete full PCDAI) or physician global assessment (PGA) compatible with quiescent disease at time of enrollment
    * No visible blood in bowel movements in the 7 days prior to enrollment
    * Normal inflammatory laboratory markers (CRP, erythrocyte sedimentation rate (ESR), Albumin in the case of PCDAI)
  * For patients with UC/IBDU:

    * Pediatric Ulcerative Colitis Activity Index (PUCAI) ≤ 20 or PGA compatible with quiescent disease
    * No visible blood in bowel movements in the 7 days prior to enrollment
* Fecal calprotectin (FC) ≥ 50 ≤ 500mcg/g or FC outside of this range but within the 20% margin of error of 500 mcg/g

Exclusion Criteria

* Positive culture for an enteropathogen up to a month prior to enrollment or during the study period.
* PCDAI >15 or sPCDAI >17.5 for patients with CD or PUCAI >20 for patients with UC or IBDU
* Presence of an ostomy or prior colonic resection
* Short bowel syndrome
* Isolated perianal disease.
* Patients requiring escalation of treatment during the intervention or preceding enrollment, defined by the following: change in dose of azathioprine/methotrexate during the preceding 12 weeks or 5-amino salicylic acid during the preceding 2 weeks, change in dosing or interval of anti-tumor necrosis factor (TNF) therapy, or any other biologic therapy (ustekinumab, vedolizumab) for the preceding infusion or injection. De-escalation of therapy (i.e stopping a medication, or spacing the interval of medication or decreasing the dose of a medication) is acceptable.
* Use of oral steroids (with the exception of budesonide) within the last 4 weeks of the screening visit or during the study period.
* Use of any antibiotics during the preceding 4 weeks or during the study period.
* Use of commercially available prebiotic preparations during the preceding 3 weeks prior to starting the study drug or during the study period.
* Non-inflammatory Crohn's disease (stricturing and/or penetrating disease behavior)
* Isolated small bowel Crohn's disease
* Previous ileocecal resection

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 51 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Alteration of gut microbiota and metabolome | 8 weeks
  The primary outcome will be assessed based on specific inulin-induced changes in microbiome composition and metabolome with a focus on short-chain fatty acid (SCFA) producers and their metabolites at week 8.

SECONDARY OUTCOMES:
Change in fecal calprotectin level | 8 weeks
  Change in fecal calprotectin following OI supplementation will be assessed 8 weeks after randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Breton, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No